CLINICAL TRIAL: NCT02128555
Title: A Randomised, Multi-centre, Non-blinded, Prospective, Parallel Group Trial of Total Ankle Replacement (TAR) Versus Ankle Arthrodesis in Patients With End Stage Ankle Osteoarthritis, Comparing Clinical Outcomes and Cost-effectiveness.
Brief Title: Total Ankle Replacement Versus Arthrodesis Trial
Acronym: TARVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/0518; 12/35/27 (Other Grant/Funding Number: NIHR HTA); ISRCTN60672307 (Registry Identifier: ISRCTN); U1111-1157-4155 (Registry Identifier: Universal Trial Number); NCT01518361 (obsolete NCT alias)
Record Dates: First submitted 2014-04-11; First posted 2014-05-01 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: ankle arthritis; osteoarthritis; total ankle replacement; arthrodesis; quality of life; musculoskeletal
MeSH Terms: conditions — Osteoarthritis; Ankylosis | interventions — Arthroplasty, Replacement, Ankle; Arthrodesis; Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthrodesis (Active Comparator): Ankle arthrodesis (fusion)
  Interventions: Procedure: Arthrodesis
- Total Ankle Replacement (Experimental): Total Ankle Replacement
  Interventions: Procedure: Total Ankle Replacement

INTERVENTIONS:
Procedure: Total Ankle Replacement — The joints are resurfaced with metal implants and a mobile plastic liner is placed between them as the gliding surface.
  Arms: Total Ankle Replacement
Procedure: Arthrodesis — The remaining damaged cartilage is removed from the ends of the bone and the two bones are then held together in compression using screws, or plates until they join to become one (bone fusion), so that there is no longer any movement at that joint.
  Other Names: Fusion
  Arms: Arthrodesis

SUMMARY:
The purpose of TARVA is to determine whether Total Ankle Replacement (TAR) provides better clinical outcomes than ankle arthrodesis in patients aged 50-85 years with end-stage ankle osteoarthritis, and compare cost-effectiveness of the two treatments

DETAILED DESCRIPTION:
This is a randomised, multi-centre, non-blinded, prospective, parallel-group trial of TAR versus ankle arthrodesis in patients with end-stage ankle osteoarthritis (OA) aged between 50 and 85 years, comparing clinical outcomes (pain-free function, quality of life (QoL), range of motion (ROM), and rate of post-procedural complications) and cost-effectiveness. TARVA is a clinician-led, pragmatic, superiority trial designed to compare the improvement in pain-free function, as assessed by the Manchester-Oxford Foot Questionnaire (MOXFQ) walking/standing domain score from pre-op to 52 weeks post-op for each surgical treatment group. A total of 328 patients will be randomly allocated on an equal basis to one of two surgical treatments: i) Total Ankle Replacement; and ii) Ankle Arthrodesis. Randomisation will be stratified by surgeon and presence of OA in two adjacent joints as determined by a pre-operative MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of end-stage ankle osteoarthritis
* Aged 50-85 years inclusive
* The surgeon believes the patient is suitable for both TAR and arthrodesis (having considered deformity, stability, bone quality, soft tissue envelope, and neurovascular status)
* The patient is able to read and understand the Patient Information Sheet (PIS) and trial procedures
* The patient is willing and able to provide written informed consent

Exclusion Criteria:

* Previous ipsilateral talonavicular, subtalar or calcaneocuboid fusion or surgery planned within 1 year of index procedure
* More than 4 lower limb joints fused (including contralateral limb, but excluding proximal interphalangeal joint fusions)
* • Unable to have MRI/CT scan (e.g. severe claustrophobia or contraindication for either scan)
* History of local bone or joint infection
* Any co-morbidity, which, in the opinion of the investigator, is severe enough to; interfere with the patient's ability to complete the study assessments or; presents an unacceptable risk to the patient's safety
* Participant in another clinical trial that would materially impact on their participation in this study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain-free function domain score | Pre-operation (baseline) to 52 weeks
  To compare the improvement in self-reported pain-free function domain score from pre-op to 52 weeks post-op for TAR versus arthrodesis, assessed by MOXFQ walking/standing domain scores.

SECONDARY OUTCOMES:
Self-reported pain-free function domain score | Pre-operation (baseline) to 26 weeks
  To compare the improvement in self-reported pain-free function domain score from pre-op to 26 weeks post-op for TAR versus arthrodesis, assessed by MOXFQ walking/standing domain scores.
Self-reported pain and social interaction domain score | Pre-operation (baseline) to 26 and 52 weeks
  To compare the improvement in self-reported pain and social interaction domain scores from pre-op to 26 and 52 weeks post-op for TAR versus arthrodesis, assessed by MOXFQ.
Self-reported physical function | Pre-operation (baseline) to 26 and 52 weeks
  To compare the improvement in self-reported physical function from pre-op to 26 and 52 weeks post-op of TAR versus arthrodesis, assessed by the Foot and Ankle Ability Measure (FAAM) questionnaire.
Self-reported quality of life | Pre-operation (baseline) to 26 and 52 weeks
  To compare the improvement in QoL from pre-op to 26 and 52 weeks post-op of TAR versus arthrodesis, assessed by EQ-5D.
Range of Motion | Pre-operation (baseline) to 52 weeks
  To compare the change in total ROM (plantarflexion and dorsiflexion) from pre-op to 52 weeks post-op of TAR versus arthrodesis, assessed by goniometer.
Adverse events | 52 weeks
  To compare the safety of TAR versus arthrodesis in terms of complications and adverse events.
Incremental cost and cost-effectiveness | 52 weeks
  To compare the incremental cost and cost-effectiveness of TAR versus arthrodesis by recording cost of all components and procedure-related costs for each surgical treatment, and using self-reported data from the Health and Social Care Services Use questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldberg, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust
Locations (17):
- United Kingdom (17):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - North Bristol NHS Trust, Bristol
  - Cardiff and Vale Orthopaedic Centre, Cardiff
  - Royal Derby Hospital, Derby
  - Royal Surrey County Hospital, Guildford
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Aintree University Hospital, Liverpool
  - Freeman Hospital, Newcastle
  - Northumbria Healthcare NHS Foundation Trust, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Northern General Hospital, Sheffield
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore
  - Wrightington Hospital, Wigan

REFERENCES:
- [Derived] Goldberg AJ, Bordea E, Chowdhury K, Hauptmannova I, Blackstone J, Brooking D, Deane EL, Bendall S, Bing A, Blundell C, Dhar S, Molloy A, Milner S, Karski M, Hepple S, Siddique M, Loveday DT, Mishra V, Cooke P, Halliwell P, Townshend D, Skene SS, Dore CJ; TARVA Study Group. Cost-Utility Analysis of Total Ankle Replacement Compared with Ankle Arthrodesis for Patients Aged 50-85 Years with End-Stage Ankle Osteoarthritis: The TARVA Study. Pharmacoecon Open. 2024 Mar;8(2):235-249. doi: 10.1007/s41669-023-00449-4. Epub 2024 Jan 8. PMID 38189868
- [Derived] Goldberg AJ, Chowdhury K, Bordea E, Blackstone J, Brooking D, Deane EL, Hauptmannova I, Cooke P, Cumbers M, Skene SS, Dore CJ. Total ankle replacement versus ankle arthrodesis for patients aged 50-85 years with end-stage ankle osteoarthritis: the TARVA RCT. Health Technol Assess. 2023 Mar;27(5):1-80. doi: 10.3310/PTYJ1146. PMID 37022932
- [Derived] Muller P, Skene SS, Chowdhury K, Cro S, Goldberg AJ, Dore CJ; TARVA Study Group. A randomised, multi-centre trial of total ankle replacement versus ankle arthrodesis in the treatment of patients with end stage ankle osteoarthritis (TARVA): statistical analysis plan. Trials. 2020 Feb 18;21(1):197. doi: 10.1186/s13063-019-3973-4. PMID 32070409
- [Derived] Goldberg AJ, Zaidi R, Thomson C, Dore CJ, Skene SS, Cro S, Round J, Molloy A, Davies M, Karski M, Kim L, Cooke P; TARVA study group. Total ankle replacement versus arthrodesis (TARVA): protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Sep 6;6(9):e012716. doi: 10.1136/bmjopen-2016-012716. PMID 27601503
- See also: TARVA website — http://www.anklearthritis.co.uk